CLINICAL TRIAL: NCT00591968
Title: Telesonography Adaptation and Use to Improve the Standard of Patient Care Within a Dominican Community
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Edward Via Virginia College of Osteopathic Medicine (Other)
Collaborators: Virginia Polytechnic Institute and State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 2007/039
Record Dates: First submitted 2007-12-31; First posted 2008-01-11 (Estimated); Last update posted 2019-07-22 (Actual); Status verified 2019-07

CONDITIONS: Ascites; Blunt Abdominal Trauma; Cholelithiasis; Cholecystitis; Cholangitis; Pancreatitis; Hydronephrosis; Abdominal Aortic Aneurysm; Hepatitis; Portal Hypertension; Urolithiasis; Abnormal Uterine Bleeding; Ovarian Mass; Ovarian Torsion
Keywords: ultrasound; telediagnosis; teleultrasound; telesonography; teleultrasonography; teleradiology; telemedicine; dominican republic; puntacana; veron; store-and-forward; asynchronous
MeSH Terms: conditions — Ascites; Cholelithiasis; Cholecystitis; Cholangitis; Pancreatitis; Hydronephrosis; Aortic Aneurysm, Abdominal; Hepatitis; Hypertension, Portal; Urolithiasis; Metrorrhagia; Ovarian Torsion | interventions — Teleradiology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (No Intervention): The control group will receive traditional ultrasound consults (i.e. travel to nearest tertiary center for intraabdominal sonographic evaluation and return with radiologist's report).
- 2 (Experimental): The experimental group will receive the teleultrasound service. Participants are randomly assigned to this group. All patients will receive a traditional clinical work-up. An ultrasound examination will be offered if, based on initial clinical evaluation by an attending physician, the patient is found to have symptoms consistent with any the following abnormalities: ascites, blunt abdominal trauma, cholelithiasis, cholecystitis, cholangitis, pancreatitis, hydronephrosis, abdominal aortic aneurysm, hepatitis, portal hypertension, urolithiasis, abnormal uterine bleeding, ovarian mass or torsion.
  Interventions: Device: SonoSite Titan portable ultrasound coupled with email telediagnosis

INTERVENTIONS:
Device: SonoSite Titan portable ultrasound coupled with email telediagnosis — Sonographic exam will be performed by principal investigator. A "first-look" diagnosis, correlated with patient symptomology and laboratory analysis, will be made at the point of care. Using a store-and-forward framework, properly formatted non-compressed sonographic images and "Request for Interpretation" (RFI) forms will be transmitted to participating radiologists. RFI forms will be used to record diagnostic findings and rate the quality of the images and/or diagnostic value using a five-point Likert scale. RFI forms will also include a five-digit patient number, age, sex, and symptomology / reason for sonographic exam. Completed RFI forms will be transmitted back to the clinic at the radiologist's earliest convenience.
  Other Names: SonoSite Titan; teleradiology; telesonography; ultrasound telediagnosis
  Arms: 2

SUMMARY:
The role of teleradiology has far reaching implications for the health of remote and underserved populations. The ability to coordinate radiographic evaluation and diagnosis from a distance has the potential to raise the standard of patient care throughout the world. Perhaps the safest and most cost effective mode of teleradiology today is telesonography. The current project attempts to determine the extent that telesonography improves the standard of care within a rural government-run primary clinic within the Dominican Republic. The work reported herein is intended to compare the use of telesonography to the current standard of sonographic examination (referral to government hospital 60km from target clinic). The study was conducted by randomly assigning 100 patients with clinical indications for sonographic examination into experimental and control groups. Following a 60-day implementation period, the following research questions will be addressed: 1) To what extent does the use of asynchronous telesonography increase the percentage of definitive diagnoses based on the total number of scans (definitive diagnoses / total number of scans)? 2) To what extent does the use of asynchronous telesonography increase the continuity of care for patients? 3) To what extent does the elapsed time between scanning and final radiological interpretation decrease with the use of asynchronous telesonography? This study will also look at the history of telemedicine / telesonography and its dissemination into the mainstream practice of medicine, explore training protocols that may be used to assist others to establish new telesonography programs in a developing nations, and discuss both advances and persistent barriers to the implementation of telesonography programs.

Hypothesis:

The use of a store-and-forward telesonography system in this setting will increase the speed and number of final diagnoses per scan received by the target clinic and will increase the continuity of care by increasing the number and speed of follow-up appointments to the target clinic.

DETAILED DESCRIPTION:
The aim of this project is comparable to the diagnostic imaging goals of the WHO including 1) make safe and reliable diagnostic imaging services available to as many as possible; 2) advise, guide and support those working in the field developing and maintaining diagnostic imaging services; 3) promote the importance of safe and appropriate diagnostic imaging services (WHO, 2007).

This project will use teleultrasound to rapidly diagnose and rule-out abdominal, retroperitoneal, and pelvic pathologies within the sole government-run ambulatory clinic of Veron, Dominican Republic. The clinic's patient records as well as the expert opinion of the clinic's physicians indicate a need for this diagnostic modality. These sources indicate a number of individuals with symptomologies suggestive of abdominal, retroperitoneal, and pelvic pathology including fever, abdominal pain, abdominal tenderness, abnormal menses, etc. (see appendix D). Given the large number of construction projects and transportation accidents within this area, it is not uncommon for individuals to present with blunt abdominal trauma. Combine these reasons and other patient indications with the clinic's remote location and the difficulty and/or resistance of members within this community to undergo timely radiological evaluation, and the utility of telesonography becomes immediately recognizable.

If the use of telesonography within this setting is shown to be feasible through this work, future projects will center on the education of native Dominican health care providers regarding the use and long-term operation of telesonography. This study could serve as a gateway to the permanent establishment of high-quality telesonography within this region of the DR. This project could also serve to augment the medical and technological knowledge of both the native health care workers and visiting U.S. medical students.

This study will contribute to the body of knowledge on telesonography by determining to what extent this technology can improve the standard of patient care within this setting. The results of this study will have implications to the practice of medicine within Veron and similar settings within the developing world. The further development of telesonography within this setting is important because it may improve the efficiency of health care through increased diagnoses, decreased time to diagnoses, and increased continuity of care.

While this pilot study focuses mainly on transabdominal evaluation of abdominal, retroperitoneal, and pelvic structures, long-term use of telesonography at the clinic could expand to include regular fetal monitoring, vascular studies, and perhaps interventional procedures granted the clinic physicians are provided with the appropriate training. Given the majority of health disparities within the DR are related to maternal, pre/perinatal, and circulatory pathologies, using telesonography to target these specific abnormalities will be the ultimate goal of a continuing telemedical presence.

ELIGIBILITY:
Inclusion Criteria:

* Clinical suspicion of one or more of the following: ascites, blunt abdominal trauma, cholelithiasis, cholecystitis, cholangitis, pancreatitis, hydronephrosis, abdominal aortic aneurysm, hepatitis, portal hypertension, urolithiasis, abnormal uterine bleeding, or ovarian mass or torsion

Exclusion Criteria:

* Urgent condition that requires immediate surgical intervention / transfer to tertiary medical center

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 106 (Actual)
Dates: Start 2008-01; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Using frequency distribution graphs, the time to final diagnosis, time to follow-up appointments, and number of successful follow-ups will be compared between the experimental and control groups. | 60 days

SECONDARY OUTCOMES:
A test for significant differences for ordinal data (Likert-scale) will be obtained using the Mann-Whitney test (if data is skewed) or the sign test (if data is non-skewed). | 60 days
Measures of variability for interval data (time) will be obtained using standard deviation. | 60 days
Measures of variability for ordinal data (Likert-scale) will be obtained using a semi-interquartile range and standard deviation. | 60 days
The measure of central tendency will be assessed using the mean. | 60 days
A number of ratios can be extracted from the data including time, number of scans, type of scan, number of reports, number of follow-ups, correct preliminary diagnoses, etc | 60 days
Correlational analysis of the interval data (time) will be obtained between groups using Spearman's rho (r2) and Pearson's r. | 60 days

CONTACTS AND LOCATIONS:
Overall Officials: James E Sutherland, D.O., Principal Investigator — Edward Via Virginia College of Osteopathic Medicine; Dean Sutphin, Ph.D., Study Chair — Edward Via Virginia College of Osteopathic Medicine
Locations (1):
- Primary Clinic of Veron, Punta Cana, La Altagracia Province, Dominican Republic